CLINICAL TRIAL: NCT01528267
Title: A Randomised, Double Blind, Sham Controlled Trial of Autologous Blood Lung Volume Reduction
Brief Title: Bronchoscopic Lung Volume Reduction Using Blood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08/H0708/100
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Emphysema
Keywords: Emphysema, lung volume reduction, autologous blood
MeSH Terms: conditions — Emphysema | interventions — Blood Transfusion, Autologous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous blood (Active Comparator): Patients will have 50mls of autologous blood injected into each of 3 bronchopulmonary segments during bronchoscopy under conscious sedation.
  Interventions: Other: Autologous blood
- Saline (Sham Comparator): Patients will have 50mls of normal saline injected into each of 3 bronchopulmonary segments during bronchoscopy under conscious sedation.
  Interventions: Other: Normal saline

INTERVENTIONS:
Other: Autologous blood — 50mls of autologous blood injected into each of 3 bronchopulmonary segments.
  Arms: Autologous blood
Other: Normal saline — 50mls of normal saline injected into each of 3 bronchopulmonary segments.
  Arms: Saline

SUMMARY:
The prupose of this study is to determine the feasibility, effectiveness, and safety of injecting blood into the airways to cause lung volume reduction in people with severe emphysema.

DETAILED DESCRIPTION:
This will be a randomised, double blind, placebo controlled trial where the response in patients treated with blood LVR will be compared to patients treated with placebo (control group). Analysis will evaluate the mean change in lobar lung volumes as determined by computed tomography (CT) scanning at 6 weeks in two study arms based on subjects' blinded bronchoscopic intervention.

Initial assessment will comprise

* Clinical evaluation
* Full pulmonary function tests (PFTs) - static and dynamic lung volumes and gas transfer
* SGRQ
* Dyspnoea Score
* CT scan

Suitable patients will then be randomised to receive either autologous blood, or normal saline injected into the target airways.

Procedures in all patients will be carried out under conscious sedation and/or anaesthesia. After bronchoscopic examination of the airways, 100ml of the patients own blood will be collected using two 50ml syringes. A balloon catheter will be inserted into the target segment and 25 mls of the blood will be injected via the balloon catheter. The balloon will be inflated and maintained in position for about 6 minutes in order to minimise the risk of overspill of blood into other areas of the lung. The balloon catheter will then be repositioned in the next segment of the target lobe of the lung and the process repeated until all the segments are treated. It is anticipated that the whole procedure will last 45-60 minutes, up to and including balloon removal.

The placebo arm will involve an identical protocol, except that injections of 30mls of 0.9% saline will replace the injections of blood. 3 segments will be 'treated'. The blood retrieved at the start of the procedure will be discarded.

A course of antibiotics or pulse of corticosteroids after the procedure will be at the discretion of the investigator. Post-operative CXRs will only be ordered if there are clinical indications (e.g. cough, fever, increased breathlessness).

Reassessment will occur at 6 weeks. This will be undertaken by a blinded assessment team with no knowledge of which study arm a patient has been randomised into, and with no access to the initial procedure record. This removes expectation and subjectivity from the assessment. Assessment will consist of the following:

* Clinical evaluation
* Full pulmonary function tests (PFTs) - static and dynamic lung volumes and gas transfer
* SGRQ
* Dyspnoea Score
* Blinding questionnaire for patient and assessment team
* CT scan

After the assessments have been completed the patients will be un-blinded and informed which treatment group they had been assigned to.

Subjects will be made aware that the process is expected to be irreversible. However, if there are any problems during the bronchoscopy (for example worsening hypoxia), then the procedure will be abandoned as soon as it is safe to do so.

A log of adverse and serious adverse events for each patient will be kept as part of the safety monitoring of the trial.

Those who are entered into the control arm of the study will be offered the real procedure at the end of the study if benefits are apparent

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Moderate to severe airflow obstruction FEV1 <50% Predicted
* Severe dyspnoea - mMRC ≥2
* Hyperinflation - total lung capacity (TLC) ≥100% predicted, RV ≥150% predicted
* Optimum COPD treatment for at least 6 weeks
* No COPD exacerbation for at least 6 weeks
* Less than 3 admissions for exacerbation in the preceding 12 months

Exclusion Criteria:

* Patient unable to provide informed consent
* Total lung CO uptake (TLCO) <15% predicted and FEV1 <15% predicted
* pO2 on air <6.0kPa
* pCO2 on air >8.0kPa
* Other major medical illness, e.g. lung cancer that will limit participation
* Clinically significant bronchiectasis
* Large bulla - more than 1/3 of hemithorax volume (i.e. where bullectomy would be more suitable) on CT scan
* Arrhythmia or cardiovascular disease that poses a risk during procedure
* Prednisolone dose greater than 10mg a day
* Prior LVRS or lobectomy
* Lung nodule requiring surgery
* Female of childbearing age with positive pregnancy test
* Subject participated in a research study of investigational drug or device in prior 30 days
* Subject taking clopidogrel, warfarin, or other anticoagulants and unable to abstain for 5 days pre-procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evidence of scarring and volume loss on CT scanning | 6 weeks

SECONDARY OUTCOMES:
To ensure no significant lung function deteriorations at 6 weeks post-procedure | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Shah, MBBS, MD, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Kobayashi H, Kanoh S. [Bronchoscopic autologous blood injection for lung volume reduction]. Nihon Kokyuki Gakkai Zasshi. 2009 Sep;47(9):765-71. Japanese. PMID 19827579